CLINICAL TRIAL: NCT05944458
Title: Efficacy of Intravenous N-Acetylcysteine in Preventing Linezolid-Induced Thrombocytopenia in Critically Ill Patients: A Double-Blind Randomized Placebo-Controlled Trial
Brief Title: Efficacy of Intravenous N-Acetylcysteine in Preventing Linezolid-Induced Thrombocytopenia in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Abdeltawab, Clinical pharmacist, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11041990
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Linezolid; Antioxidant; Thrombocytopenia; Critical Illness; ICU
MeSH Terms: conditions — Thrombocytopenia; Critical Illness | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine group (Active Comparator): Generic name: N-acetylcysteine.
  * Trade name: Fluimucil.
  * Company: Zambon.
  * Dosage form: ampoules for intravenous administration.
  * Dose: 600mg taken every 12 hours daily with a fixed dose as there is no need for renal or hepatic adjustment, starting with the inception of linezolid therapy.
  * Duration: for 14 days post linezolid discontinuation or until ICU discharge, whichever came first.
  Interventions: Drug: N acetyl cysteine
- Standard of care (Placebo Comparator): They will receive standard of care (Platelets monitoring daily, linezolid discontinuation if platelet count less than 50000 or clinically appropriate and platelet transfusion according to the institutional protocol) plus placebo (20 ml normal saline twice daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N acetyl cysteine — Fluimucil 600 mg iv to be taken twice daily as infusion
  Other Names: Fluimucil; NAC
  Arms: N-acetylcysteine group
Drug: Placebo — 20 ml normal saline iv every 12 hours
  Arms: Standard of care

SUMMARY:
* Study the effect of acetylcysteine on decreasing the incidence of LIT in critically ill patients.
* Study the impact of acetylcysteine on the time to onset of LIT and the time to recovery of platelets.

DETAILED DESCRIPTION:
Primary outcome: difference in incidence of LIT between patients who received NAC and patients who didn't.

* Primary outcome definition: Defined as platelets < 150000 OR decrease > 50% of baseline platelets.
* Secondary outcome: difference in Time to onset of LIT and time to recovery between the 2 groups. Blood products transfusion, bleeding, length of stay, and in-hospital mortality incidence between 2 groups.
* Secondary outcome definitions: after having thrombocytopenia, regardless of discontinuation of linezolid, recovery is defined as the restoration and maintenance of platelet counts > 70% of baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Admitted to the Intensive Care Unit (ICU)
* Candidates for intravenous linezolid therapy for ≥ 48 hours

Exclusion Criteria:

* Baseline platelet count < 50 × 10⁹/L
* Diagnosis of malignancy
* Receipt of any chemotherapeutic agent within the past 6 months
* Positive COVID-19 RT-PCR test at admission
* Diagnosis of immune thrombocytopenia
* Presence of splenomegaly
* Presence of liver cirrhosis
* Presence of hepatitis C
* Refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
difference in incidence of LIT between patients who received NAC and patients who didn't. | From starting linezolid untill 14 days after linezolid discontinuation or ICU discharge whichever comes first.
  Defined as platelets < 150000 OR decrease > or = 50% of baseline platelets.

SECONDARY OUTCOMES:
Blood products transfusion, bleeding, length of ICU stay, and in-ICU mortality incidence between 2 groups. | From start linezolid until ICU discharge
Difference in time to platelet recovery between the 2 groups | From thrombocytopenia onset to recovery, assesed up to 14 days after linezolid discontinuation or ICU discharge whichever comes first
  after having thrombocytopenia, regardless of discontinuation of linezolid, recovery is defined as the restoration and maintenance of platelet counts > 70% of baseline values
Difference in time to thrombocytopenia onset between the 2 groups | From linezolid start date until date of first thrombocytopenia event, assessed up to 14 days after linezolid discontinuation or ICU discharge whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdeltawab, Pharm D, Principal Investigator — Clinical pharmacy, 15 May hospital
Locations (1):
- 15 May hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdeltawab M, Ebid AH, Ahmed O, Mobarez MA, Ibrahim M. N-acetylcysteine reduces incidence and duration of linezolid-associated thrombocytopenia in critically ill patients: A randomized controlled trial. Environ Toxicol Pharmacol. 2026 Jan 21;122:104944. doi: 10.1016/j.etap.2026.104944. Online ahead of print. PMID 41577060